CLINICAL TRIAL: NCT05642702
Title: Evaluation of Dermatological Safety of Test Products by 24 Hours Patch Test Under Complete Occlusion or Semi Occlusion or Open Patch on Adult Healthy Human Subjects
Brief Title: Primary Irritation Patch Test (PIPT) Study Conducted at NovoBliss Research for Shared Panel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Nanobrid Innovations Private Limited (Industry)
Responsible Party: Principal Investigator, Dr Nayan Patel, Principal Investigator, NovoBliss Research Pvt Ltd
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NBSP22-PIPT; NBSP22-PIPT-0030-NI (Other: NovoBliss Research Private Limited)
Record Dates: First submitted 2022-11-12; First posted 2022-12-08 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Healthy
MeSH Terms: interventions — Ascorbic Acid; Niacinamide; long-chain-aldehyde dehydrogenase; Solutions; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Evaluator Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Test Product Code A (Experimental): Peptide complexed HA Age Defying Gel with Vitamin C & Niacinamide -
  Interventions: Other: Peptide complexed HA Age Defying Gel with Vitamin C & Niacinamide
- Test Product Code B (Experimental): Peptide complexed HA Age Defying Gel with Natural Extracts
  Interventions: Other: Peptide complexed HA Age Defying Gel with Natural Extracts
- Test Product Code C (Experimental): Peptide complexed HA Age Defying Gel with Vitamin C & Natural Extracts
  Interventions: Other: Peptide complexed HA Age Defying Gel with Vitamin C & Natural Extracts
- Positive Control (Active Comparator): Sodium Lauryl Sulphate (SLS) analytical grade 1 % w/v
  Interventions: Other: 1% w/v Sodium Lauryl Sulphate (SLS) solution
- Negative Control (Active Comparator): Sodium chloride (Isotonic Saline Solution) Injection IP 0.9 % w/v
  Interventions: Other: Sodium chloride (Isotonic Saline Solution) Injection IP 0.9 % w/v

INTERVENTIONS:
Other: Peptide complexed HA Age Defying Gel with Vitamin C & Niacinamide — Semi Solid, Hydrophilic - Gel, A 0.04 mL of test sample will be dispensed onto the center of an appropriately sized filter paper will be placed in the designated IQ/Finn chambers prefixed to a micropore tape.
  Other Names: Skin Care product
  Arms: Test Product Code A
Other: Peptide complexed HA Age Defying Gel with Natural Extracts — Semi Solid, Hydrophilic - Gel, A 0.04 mL of test sample will be dispensed onto the center of an appropriately sized filter paper will be placed in the designated IQ/Finn chambers prefixed to a micropore tape.
  Other Names: Skin Care product
  Arms: Test Product Code B
Other: Peptide complexed HA Age Defying Gel with Vitamin C & Natural Extracts — Semi Solid, Hydrophilic - Gel, A 0.04 mL of test sample will be dispensed onto the center of an appropriately sized filter paper will be placed in the designated IQ/Finn chambers prefixed to a micropore tape.
  Other Names: Skin Care product
  Arms: Test Product Code C
Other: 1% w/v Sodium Lauryl Sulphate (SLS) solution — 1g of Sodium Lauryl Sulphate will be dissolved in distilled water and made up to 100 mL solution using distilled water. A 0.04 mL of test sample will be dispensed onto the center of an appropriately sized filter paper will be placed in the designated IQ/Finn chambers prefixed to a micropore tape.
  Other Names: Positive Control
  Arms: Positive Control
Other: Sodium chloride (Isotonic Saline Solution) Injection IP 0.9 % w/v — A 0.04 mL of 0.9% w/v solution of Isotonic Saline Solution will be dispensed on the center of an appropriately sized filter paper, which will be further placed in the designated IQ/Finn chambers prefixed to a micropore tape.
  Other Names: Negative Control
  Arms: Negative Control

SUMMARY:
This is a single-center, evaluator-blinded study in healthy adult human subjects. Single 24-hour application of sponsor(s) provided test products along with positive and negative controls will be kept in contact with the skin of subjects under occlusion for at least 24 hours (+ 2 hours). The study can be conducted in a single group. Safety will be assessed throughout the study by monitoring adverse events.

The subject's back between the scapula and waist will be utilized as application sites. Application sites will be evaluated for scoring the reaction, namely, erythema, dryness, and wrinkles on a 0-4 point scale separately for each parameter and edema on another 0-4 points scale as per the Draize Scale after 30+5 minutes of patch removal, 24±2 hours and 168±2 hours after patch removal.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the dermatological safety of the test products by 24 Hours patch test under complete occlusion on healthy adult human subjects and adequate representation of varied skin types (Oily, Dry, Normal, and Combination).

This is a single-center, evaluator-blinded study in healthy adult human subjects. Single 24-hour application of sponsor(s) provided test products along with positive and negative controls will be kept in contact with the skin of subjects under occlusion for at least 24 hours (+ 2 hours). The study can be conducted in a single group. Safety will be assessed throughout the study by monitoring adverse events. The subject's back i.e. between the scapula and waist will be utilized as application sites.

26 subjects with varied skin types (Oily, Dry, Normal, and Combination, preferably equal ratio) will be enrolled in the study to get 24 completed subjects at the end of study.

The expected total study duration will be approximately 9 days from patch application day.

The duration of this study will be 9 days from enrollment day. There are total of 3 visits in this study and one optional visit.

* Visit 01: Screening, Enrollment, and Patch Application (Day 01)
* Visit 02: Patch Removal after 24 hours of application & 30 + 5 min Irritation scoring upon patch removal (Day 02)
* Visit 03: 24 (± 2) hours Irritation Scoring (Day 03) after patch removal
* Visit 04: The subject will be contacted telephonically on Day 08 for any signs of irritation at the patch application site. Follow-up visit for reactions if any to confirm recovery (Optional, if deemed necessary) [Irritation scoring at 168±2 hours post-patch removal (Day 09)].

Application Sites (Back) will be evaluated for scoring the reaction, namely, erythema, dryness, wrinkles on a 0-4 point scale separately for each parameter and oedema on another 0-4 points scale as per the Draize Scale after 30 + 5 minutes of patch removal (Day 02), 24±2 hours (Day 03) and 168±2 hours (Day 09) after the patch removal.

Scoring data will be updated in tabular format and mean irritation scoring will be obtained from irritation scores and the same will be included in the final Product Summary Report for all test products after completion of the study.

Demographic characteristics and results of the study will be summarized. Any AEs will be summarized with a number and a percentage.

Four parameters namely erythema, dryness, wrinkles and oedema will be scored separately on the irritation scoring sheet. Irritation scoring data will be updated in tabular format. Data of each subject that has completed the initial 03 study visits i.e. Day 01, Day 02, and Day 03 of the study will be considered for Mean Irritation Score Derivation. Mean Irritation Score (MIS) and standard deviation will be calculated using a standard statistical formula for each product. The Product irritancy level will be classified and reported based on the classification of Mean Irritation Score per sec#17.1. Standard deviation will be calculated to provide variability of data.

For calculation of Mean Irritation Score of erythema, dryness and wrinkles the highest score will be taken.

MIS = Total score (highest score from Erythema, dryness, wrinkles + Oedema) for each test product / Total no. of Subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years (both inclusive) at the time of consent.
2. Sex: Males and non-pregnant/non-lactating females (preferably equal number of males and females).
3. Subject with normal Fitzpatrick skin type III to V (Human skin colour determination scale).
4. Females of childbearing potential must have a negative urine pregnancy test performed on Day 01 prior to patch application.
5. Subject who do not have any previous history of adverse skin conditions and are not under any medication likely to interfere with the results.
6. Subject is in good general health as determined by the Investigator on the basis of medical history.
7. Subjects is willing to maintain the test patches in designated positions for 24 Hours.
8. Subject is willing and able to follow the study directions, to participate in the study, returning for all specified visits.
9. Subject must be able to understand and provide written informed consent to participate in the study.
10. Subject is willing to refrain from vigorous physical exercise during the study period and follow all the instruction given.

Exclusion Criteria:

1. Subject having skin irritation, blemishes, excessive hair, moles, pigmentation, pimples, marks (e.g. tattoos (within the previous 3 months), scars, sunburn), open wounds, cuts, abrasions, irritation symptoms or any dermatological condition on the test site(s) i.e. back that can interfere with the reading.
2. Medication which may affect skin response and/or past medical history.
3. Subject having history of diabetes
4. Subject have history of mastectomy for cancer involving removal of lymph nodes within the past year, or treatment of any type of cancer within the last 6 months.
5. Subject suffering from any active clinically significant skin diseases which may contraindicate.
6. Subject having history of any skin diseases including eczema, atopic dermatitis or active cancer.
7. Participation in any patch test for irritation or sensitization within the last four weeks.
8. Subject having history of asthma or COPD (Chronic obstructive pulmonary disease).
9. Use of any:

   i. Prescribed or over-the-counter (OTC) anti-inflammatory drug within five (5) days prior to application.

   ii. Antihistamine medication or immunosuppressive drugs within seven (7) days prior to first patch application.

   iii. Systemic or topical corticosteroids at patch site within four (4) weeks of test product application (steroidal nose drops and/or eye drops are permitted)
10. Topical drugs used at application site.
11. Subject with Self-reported Immunological disorders such as HIV positive, AIDS and/or systemic lupus erythematous.
12. Individual who has a medical condition or is taking or has taken a medication which, in the Investigator's judgment, makes the subject ineligible or places the subject at undue risk.
13. Subject with known allergy or sensitization to medical adhesives, bandages.
14. Participation in other patch study simultaneously.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-12-05 (Estimated); Primary Completion 2022-12-13 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Change from Irritation Potential of the test product from Baseline to Post application | Irritation Scoring at 30 minutes, and 24 hours, 168 hours post patch removal.
  To evaluate the dermatological irritation potential of the test products by applying Patch Test Under Complete Occlusion for continuous 24 Hours exposure on healthy adult human subjects and adequate representation of varied skin types (Oily, Dry, Normal and Combination)

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | At 30 minutes (on Day2) and 24 hours (on Day 3) post patch removal and up to 9 days from the Day 1.
  Incidence of Treatment-Emergent Adverse Events regarding acute strong dermal reactions such as dryness, swelling, redness, scaling reported, during the clinical conduct on Day1, 2, 3 and day 7 post patch removal and entire study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nayan K Patel, MBBS, Principal Investigator — Medical Director

IPD SHARING:
Plan to Share IPD: No